CLINICAL TRIAL: NCT06393530
Title: Erector Spinae Plane Block for Cervical Spine Surgery. A Prospective, Randomized, Double-blinded Clinical Trial.
Brief Title: Erector Spinae Plane Block for Cervical Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 545/23
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Spine Fusion; Spine Disease; Spinal Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham group (Sham Comparator): Bilateral ESPB under ultrasound guidance (adjusted to the incision line): 2 x 20ml/kg 0,9% normal saline
  Interventions: Drug: 0.9%sodium chloride
- ESPB group (Active Comparator): Bilateral ESPB under ultrasound guidance (adjusted to the incision line): 2 x 20ml/kg 0.2% Ropivacaine
  Interventions: Drug: 0.2% ropivacaine

INTERVENTIONS:
Drug: 0.9%sodium chloride — Bilateral ESPB under ultrasound guidance (adjusted to the incision line): 2 x 20ml/kg 0,9% normal saline
  Other Names: 0,9% normal saline
  Arms: Sham group
Drug: 0.2% ropivacaine — Bilateral ESPB under ultrasound guidance (adjusted to the incision line): 2 x 20ml/kg 0,2% ropivacaine
  Other Names: 0,2% ropivacaine
  Arms: ESPB group

SUMMARY:
The study aims to assess the interfacial plane blocks' effect on pain level, course of postoperative rehabilitation, and anti-inflammatory analgesic effect.

DETAILED DESCRIPTION:
This study evaluates the analgesic efficacy in adults of bilevel, bilateral erector spinae plane (ESP) blocks after posterior cervical spinal fusion surgery by assessing postoperative pain scores and opiate requirements as the primary outcome measures. We aim to investigate how ESP blocks, performed under ultrasound guidance at the two vertebral levels, contribute to postoperative pain control. This will be determined by measuring numerical rating pain scores repeatedly following surgery and opiate consumption until the patient is discharged from the hospital. These primary outcome measures will be compared between a treatment group of participants receiving ESP blocks and a control group receiving a sham block. Our primary hypothesis is that ESP blocks significantly reduce postoperative pain and opiate requirements.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary posterior cervical decompression and stabilization with instrumentation involving multi-levels in the cervical region,
* aged >18 years and <100 years
* ASA physical status 1, 2 or 3.

Exclusion Criteria:

* refuse to participate,
* history of opioid abuse,
* infection of the puncture site,
* aged <18 years and >100 years
* ASA 4 and 5

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-17 (Actual)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 16 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 20 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 36 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
NLR | 12 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 12 hours after surgery
  Platet-to-lymphocyte ratio
PLR | 24 hours after surgery
  Platet-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platet-to-lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Domagalska, Ph.D., Study Chair — Poznań University of Medical Science
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No